CLINICAL TRIAL: NCT06335524
Title: Infant-Maternal Partnership and Cognitive Training Study for Preterm Infants: A Randomized Clinical Trial
Brief Title: Infant-Maternal Partnership and Cognitive Training Study for Preterm Infants
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300012718; UAB (Other: UAB)
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Child Development; Infant Development; Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver-implemented early developmental intervention (EDI) using finger puppets (Experimental): Caregivers of infants in the intervention group will receive finger-puppets and additional training pertaining to infant parent interaction and developmentally appropriate infant communication training.
  Interventions: Behavioral: Finger puppet; Behavioral: Bookworm reading intervention training and routine EDI care.
- Routine EDI care including Bookworm training (Active Comparator): All study participants will receive Bookworm reading intervention training and routine EDI care.
  Interventions: Behavioral: Bookworm reading intervention training and routine EDI care.

INTERVENTIONS:
Behavioral: Finger puppet — The intervention group will receive finger-puppets and additional training pertaining to infant parent interaction and developmentally appropriate infant communication training.
  Arms: Caregiver-implemented early developmental intervention (EDI) using finger puppets
Behavioral: Bookworm reading intervention training and routine EDI care. — Routine EDI care including Bookworm training.

SUMMARY:
This study will test the hypothesis that in preterm infants a caregiver-implemented early developmental intervention (EDI) using finger puppets to develop joint attention and encourage interactive communication with routine EDI care including Bookworm training compared with routine EDI care including Bookworm training alone will increase the Ages and Stages Questionnaire® score at 12 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* inborn at UAB, delivered at less than 34 weeks' gestation, 32-39 weeks' PMA, off sedatives, and off invasive respiratory support.

Exclusion Criteria:

* a major malformation, a known syndrome, enrolled in a competing trial targeting neurodevelopmental outcomes as a primary outcome.

Ages: 1 Week to 17 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
ASQ-3 scores | 12 months corrected age
  Ages and Stages Questionnaires 3rd Edition

SECONDARY OUTCOMES:
ASQ-3 scores | 24 months corrected age
  Ages and Stages Questionnaires 3rd Edition
ASQ scores below -2SD | 12 months corrected age
  Ages and Stages Questionnaires 3rd Edition
ASQ scores below -2SD | 24 months corrected age
  Ages and Stages Questionnaires 3rd Edition
ASQ scores below -1SD | 12 months corrected age
  Ages and Stages Questionnaires 3rd Edition
ASQ scores below -1SD | 24 months corrected age
  Ages and Stages Questionnaires 3rd Edition
ASQ-SE2 scores | 12 months corrected age
  Ages and Stages Questionnaires 3rd Edition
ASQ-SE2 scores | 24 months corrected age
  Ages and Stages Questionnaires 3rd Edition
Severe neurodevelopmental impairment | 24 months corrected age
  Composite outcome based on BSID scores, GMFCS, Vision, Hearing
Moderate or severe neurodevelopmental impairment | 24 months corrected age
  Composite outcome based on BSID-IV scores, GMFCS, Vision, Hearing
Cognitive Composite Score on BSID-IV | 24 months corrected age
  Bayley's Scales of Infant Development IV cognitive composite score
Language Composite Score on BSID-IV | 24 months corrected age
  Bayley's Scales of Infant Development IV language composite score
Motor Composite Score on BSID-IV | 24 months corrected age
  Bayley's Scales of Infant Development IV motor composite score
Edinburgh Postnatal Depression Scale | 6 months
  Maternal scores on Edinburgh Postnatal Depression Scale
MCHAT score | 24 months corrected age
  Modified Checklist for Autism in Toddlers

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No